CLINICAL TRIAL: NCT02129673
Title: A Phase 1/2 Multicenter, Randomized, Controlled Dose-Finding Study to Evaluate the Safety and Ocular Hypotensive Efficacy of 3 Dose Levels of the VS101 Subconjunctival Latanoprost Insert for 3 Months in Subjects With Open-Angle Glaucoma or Ocular Hypertension
Brief Title: A Phase 1/2 Multicenter, Randomized, Study to Evaluate the Safety and Efficacy of VS101 Subconjunctival Latanoprost Insert in Subjects With Open-Angle Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ViSci Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VS101-CS201
Record Dates: First submitted 2014-04-30; First posted 2014-05-02 (Estimated); Last update posted 2018-03-14 (Actual); Status verified 2017-10

CONDITIONS: Open Angle Glaucoma; Ocular Hypertension
Keywords: Glaucoma; Intra-ocular pressure; Slow Release; Controlled release
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension; Glaucoma | interventions — Latanoprost; Ophthalmic Solutions

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- VS101 Insert Dose A (Experimental): VS101 Insert Dose A placed under the conjunctiva
  Interventions: Drug: VS101 Insert Dose A
- VS101 Insert Dose B (Experimental): VS101 Insert Dose B placed under the conjunctiva
  Interventions: Drug: VS101 Insert Dose B
- VS101 Insert Dose C (Experimental): VS101 Insert Dose C placed under the conjunctiva
  Interventions: Drug: VS101 Insert Dose C
- Latanoprost 0.005% eye drops (Active Comparator): Latanoprost 0.005% eye drops administered once daily on the eye
  Interventions: Drug: Latanoprost 0.005% eye drops

INTERVENTIONS:
Drug: VS101 Insert Dose A — Sustained release of latanoprost into the eye
  Arms: VS101 Insert Dose A
Drug: VS101 Insert Dose B — Sustained release of latanoprost into the eye
  Arms: VS101 Insert Dose B
Drug: VS101 Insert Dose C — Sustained release of latanoprost into the eye
  Arms: VS101 Insert Dose C
Drug: Latanoprost 0.005% eye drops — Latanoprost 0.005% eye drops administered once daily on the eye
  Arms: Latanoprost 0.005% eye drops

SUMMARY:
Slow release formulation of latanoprost is compared for safety and pressure-lowering efficacy with topically administration of commercially available latanoprost in patient with glaucoma and ocular hypertension

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Open angle glaucoma or Ocular Hypertension

Exclusion Criteria:

* uncontrolled medical conditions
* wearing of contact lenses

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2014-05; Primary Completion 2017-05 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Intra-ocular pressure | 12 weeks

SECONDARY OUTCOMES:
Intra-ocular pressure | Week 8
Intra-ocular pressure | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Speciality Eyecare Centre, Bellevue, Washington, United States